CLINICAL TRIAL: NCT02035891
Title: Low-dose Colchicine Intervention in Patients With Type 2 Diabetes Mellitus and Microalbuminuria: Chongqing Study
Brief Title: Low-dose Colchicine in Patients With Type 2 Diabetes Mellitus and Microalbuminuria
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qifu Li, director of the Endocrinology Department, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQMU-2013-QLi
Record Dates: First submitted 2014-01-04; First posted 2014-01-14 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Diabetic Nephropathy
Keywords: colchicine; urinary albumin-to-creatinine ratio; carotid Intima-Media Thickness; overt nephropathy; Type 2 diabetes
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2 | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- colchicine (Active Comparator): 0.5mg/d colchicine
  Interventions: Drug: colchicine 0.5mg/d
- placebo (Placebo Comparator): appearance is same as colchicine
  Interventions: Drug: placebo 0.5mg/d

INTERVENTIONS:
Drug: colchicine 0.5mg/d — on the basis of standard therapy to manage hyperglycemia, hypertension,dislipidemia etc.
  Arms: colchicine
Drug: placebo 0.5mg/d — on the basis of standard therapy to manage hyperglycemia, hypertension,dislipidemia etc.
  Arms: placebo

SUMMARY:
1. The primary objective of this study was： in patients with type 2 diabetes and microalbuminuria who have been receiving stable treatment of angiotensin-converting enzyme inhibitor/angiotensin II receptor blocker (ACEI/ARB) for at least 3 months, whether low-dose colchicine slows the progression of microvascular complications.
2. The secondary objective of this study was： (1) whether low-dose colchicine could reduce Urinary Albumin To Creatinine Ratio (UACR), or improve eGFR in patients with type 2 diabetes and microalbuminuria; (2) whether low-dose colchicine decreases carotid intima-media thickness(IMT) in patients with type 2 diabetes and microalbuminuria; (3) whether low-dose colchicine reduces the risk of cardiovascular events or mortality in patients with type 2 diabetes and microalbuminuria.

DETAILED DESCRIPTION:
BACKGROUND-Previous study reported that colchicine 0.5 mg/day, in addition to statins and other standard secondary prevention therapies, was effective for the prevention of cardiovascular events in patients with stable coronary disease. An experiment conducted by Li et al. showed that twenty-four-hour urinary albumin excretion was reduced after 6 months colchicine treatment in rats with diabetic nephropathy.As both micro and macrovascular complications of diabetes are closely associated with inflammation,with the anti-inflammation property,colchicine might reduce risk for micro and macrovascular complications of diabetes.

STUDY DESIGN-Patients with type 2 diabetes and microalbuminuria(30mg/g Cr≤UACR≤300mg/g Cr) who have received stable dosage of ACEI/ARB for at least 3 months will be randomized to receive colchicine 0.5 mg/day or placebo.

This trial includes four phases:

* Phases 1: A prospective, randomized，double-blind, control study, aims at evaluating microvascular events from date of randomization until the third year. Other parameters included evaluating changes of UACR, eGFR, CIMT from baseline to the follow-up.
* Phases 2: A prospective observational study, aims at evaluating macrovascular and microvascular events from date of randomization until the 6th year.

SAFETY AND DATA MANAGEMENT-Independent Safety and Data Monitoring Committee has been set up to monitor the safety and tolerability of the subjects; this committee will analyze data independent of investigators at the end of any one phase.

ELIGIBILITY:
Inclusion Criteria:

* Well informed of the procedures of this trial and informed consent is obtained
* Voluntarily accept standardized treatment
* 30-70 years old, gender is not limited
* Diagnosed as type 2 diabetes and have received standardized hypoglycemic therapy
* Have been receiving stable doses of ACEI or ARBs for at least 3 months
* Two of three examinations of UACR at random urine are 30-300 mg/g Cr (infection or other factors were ruled out) in 3 months
* Well compliance
* Capable of self blood Glucose monitoring

Exclusion Criteria:

* Pregnant or lactating
* Type 1 diabetes
* Poor blood glucose control（HbA1c>11%）
* A history of malignant tumor
* Abnormal liver or renal function (defined as alanine aminotransferase(ALT)>2.5 times higher than normal range,or eGFR<30 mL/min per 1•73 m²)
* Poor blood pressure control [systolic blood pressure(SBP)>180mmHg,or diastolic blood pressure(DBP)>110mmHg]
* With severe heart disease,cardiac function worse than grade II,anemia(Hb<9.0g/d1)
* Continuous use of colchicine or non-steroidal anti-inflammatory drugs (except aspirin) more than one week in recent 3 months
* History of gout
* Blood routine test indicates that the white blood cell count(WBC) <3*109/l
* Body Mass Index(BMI)<18.5 or ≥35kg/m2
* Drug or alcohol abuse
* Accompanying mental disorder who can't collaborate
* Abnormal digestion and absorption function
* Other endocrine diseases
* Other chronic diseases needed long-term glucocorticoid treatment
* With severe infection, immune dysfunction
* A history of colchicine allergies or allergic constitution

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
The incidence of overt nephropathy | 3 years
  overt nephropathy is defined as any one of the events described below: （1） UACR greater than 300 mg/g Cr; (2) 24 h urinary albumin greater than 300 mg; (3)doubling of the serum creatinine level to at least 200 μmol per liter; (4)the need for renal-replacement therapy;(5) death due to renal disease.

SECONDARY OUTCOMES:
The proportion of patients achieving at least a 15% reduction in UACR | 3 years
  Renal outcome
Changes in estimated Glomerular Filtration Rate (eGFR) | 3 years
  Renal outcome
The number of patients who have new or worsening diabetic neuropathy | 3 years
  diabetic neuropathy was assessed based on biothesiometer.
The number of patients who have new or worsening diabetic retinopathy | 3 years
  Diabetic retinopathy was diagnosed according to the six-level grading scale of the European Community- funded Concerted Action Programme into the Epidemiology and Prevention of Diabetes (EURODIAB)
changes in CIMT from baseline to the 3rd year | 18 months and 3 year
  cardiovascular outcome
The number of patients who have new cardiovascular events | 6 years
  cardiovascular events include death from cardiovascular causes, nonfatal stroke, nonfatal myocardial infarction, coronary-artery bypass grafting, percutaneous coronary intervention or revascularization for peripheral atherosclerotic arterial disease, and amputation because of ischemia
changes of UACR | 6 years
  evaluated at 6, 12, 18, 24, 36, 48, 60, 72 months
changes of eGFR | 6 years
  evaluated at 6, 12, 18, 24, 36, 48, 60, 72 months
Death from any cause | 6 years
  All-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Qifu Li, PhD, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Nidorf SM, Eikelboom JW, Budgeon CA, Thompson PL. Low-dose colchicine for secondary prevention of cardiovascular disease. J Am Coll Cardiol. 2013 Jan 29;61(4):404-410. doi: 10.1016/j.jacc.2012.10.027. Epub 2012 Dec 19. PMID 23265346
- [Background] Nidorf M, Thompson PL. Effect of colchicine (0.5 mg twice daily) on high-sensitivity C-reactive protein independent of aspirin and atorvastatin in patients with stable coronary artery disease. Am J Cardiol. 2007 Mar 15;99(6):805-7. doi: 10.1016/j.amjcard.2006.10.039. Epub 2007 Jan 16. PMID 17350370
- [Background] Navarro-Gonzalez JF, Mora-Fernandez C, Muros de Fuentes M, Garcia-Perez J. Inflammatory molecules and pathways in the pathogenesis of diabetic nephropathy. Nat Rev Nephrol. 2011 Jun;7(6):327-40. doi: 10.1038/nrneph.2011.51. Epub 2011 May 3. PMID 21537349
- [Background] Bots ML, Visseren FL, Evans GW, Riley WA, Revkin JH, Tegeler CH, Shear CL, Duggan WT, Vicari RM, Grobbee DE, Kastelein JJ; RADIANCE 2 Investigators. Torcetrapib and carotid intima-media thickness in mixed dyslipidaemia (RADIANCE 2 study): a randomised, double-blind trial. Lancet. 2007 Jul 14;370(9582):153-160. doi: 10.1016/S0140-6736(07)61088-5. PMID 17630038
- [Background] de Zeeuw D, Agarwal R, Amdahl M, Audhya P, Coyne D, Garimella T, Parving HH, Pritchett Y, Remuzzi G, Ritz E, Andress D. Selective vitamin D receptor activation with paricalcitol for reduction of albuminuria in patients with type 2 diabetes (VITAL study): a randomised controlled trial. Lancet. 2010 Nov 6;376(9752):1543-51. doi: 10.1016/S0140-6736(10)61032-X. PMID 21055801
- [Background] ADVANCE Collaborative Group; Patel A, MacMahon S, Chalmers J, Neal B, Billot L, Woodward M, Marre M, Cooper M, Glasziou P, Grobbee D, Hamet P, Harrap S, Heller S, Liu L, Mancia G, Mogensen CE, Pan C, Poulter N, Rodgers A, Williams B, Bompoint S, de Galan BE, Joshi R, Travert F. Intensive blood glucose control and vascular outcomes in patients with type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2560-72. doi: 10.1056/NEJMoa0802987. Epub 2008 Jun 6. PMID 18539916
- [Background] Gaede P, Vedel P, Parving HH, Pedersen O. Intensified multifactorial intervention in patients with type 2 diabetes mellitus and microalbuminuria: the Steno type 2 randomised study. Lancet. 1999 Feb 20;353(9153):617-22. doi: 10.1016/S0140-6736(98)07368-1. PMID 10030326
- [Background] ORIGIN Trial Investigators; Gerstein HC, Bosch J, Dagenais GR, Diaz R, Jung H, Maggioni AP, Pogue J, Probstfield J, Ramachandran A, Riddle MC, Ryden LE, Yusuf S. Basal insulin and cardiovascular and other outcomes in dysglycemia. N Engl J Med. 2012 Jul 26;367(4):319-28. doi: 10.1056/NEJMoa1203858. Epub 2012 Jun 11. PMID 22686416
- [Background] Li JJ, Lee SH, Kim DK, Jin R, Jung DS, Kwak SJ, Kim SH, Han SH, Lee JE, Moon SJ, Ryu DR, Yoo TH, Han DS, Kang SW. Colchicine attenuates inflammatory cell infiltration and extracellular matrix accumulation in diabetic nephropathy. Am J Physiol Renal Physiol. 2009 Jul;297(1):F200-9. doi: 10.1152/ajprenal.90649.2008. Epub 2009 Apr 15. PMID 19369290